CLINICAL TRIAL: NCT02505893
Title: A Monocentric, Open-label Pilot Study to Assess the Safety and Efficacy of Minimal Islet Transplantation in Patients With New-onset Type 1 Diabetes
Brief Title: Minimal Islet Transplant at Diabetes Onset
Acronym: MITO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Collaborators: Italian Diabetes Foundation (Other)
Responsible Party: Principal Investigator, Lorenzo Piemonti, Deputy Director Diabetes Researh Institute, Ospedale San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRI-MITO 1/2014
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sirolimus

ARMS (1):
- Treated (Experimental): The investigational treatment will be islet transplant in the presence of induction with ATG/G-CSF and rapamycin treatment for one month. One thousand and five hundred (1,500) equivalent islet for Kg of body weight, isolated from a single brain-dead donor, will be infused into the patient's liver. ATG will be administered IV (central vein) at a total dose of 6 mg/kg up to day 6 post-transplant. Pegylated G-CSF (6 mg/dose) will be administered SC every 2 weeks for 6 doses (12 weeks) beginning after the last ATG infusion. Rapamycin will be administered orally at a starting dose of 0.2 mg/kg once a day, then targeted to blood trough level of 8-10 ng/mL and suspended one month after transplant.
  Interventions: Biological: Human pancreatic islet; Drug: ATG; Drug: Pegylated G-CSF; Drug: Rapamycin

INTERVENTIONS:
Biological: Human pancreatic islet — One thousand and five hundred (1,500) equivalent islet for Kg of body weight, isolated from a single brain-dead donor, will be infused into the patient's liver.
Drug: ATG — ATG will be administered IV (central vein) at a total dose of 6 mg/kg up to day 6 post-transplant
Drug: Pegylated G-CSF — Pegylated G-CSF (6 mg/dose) will be administered SC every 2 weeks for 6 doses (12 weeks) beginning after the last ATG infusion
Drug: Rapamycin — Rapamycin will be administered orally at a starting dose of 0.2 mg/kg once a day, then targeted to blood trough level of 8-10 ng/mL and suspended one month after transplant.

SUMMARY:
This is a prospective phase 2, single-arm, mono-center pilot study. It has been designed to investigate whether giving the combination therapy consisting of minimal islet transplantation (1500 EIQ/Kg body weight), Thymoglobulin® (ATG), Rapamune® (rapamycin) and Neulasta® (pegfilgastrim) to patients with Type 1 Diabetes (T1D) at onset is safe and secondarily, if it will preserve insulin production. It will involve 6 patients with new-onset T1D. Each patient will be involved in the study for a screening period and a post-islet transplantation study period of 52±2 weeks, to include 1 treatment cycles of 12 weeks, assessment during treatment and 5 follow-up visits scheduled at weeks 2±1 (14 days), 4±1 (month 1), 12±2 (month 3), 26±2 (month 6) and 52±2 (month 12).

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Mentally stable and able to comply with the protocol procedures for the duration of the study, including scheduled follow-up visits and examinations
* New-onset T1D (diagnosis of diabetes within 180 days prior to enrolment). Documentation of the diagnosis of T1DM (and not just insulin deficiency), including the date of diagnosis, must be obtained from the diagnosing physician.
* Residual beta-cell function (fasting C-peptide >0.3 ng/mLwhen plasma glucose level is > 70 mg/dL and ≤ 200 mg/dL.
* Positive for at least one of the following autoantibodies typically associated with T1DM: antibody to glutamic acid decarboxylase (anti-GAD) antibody to protein tyrosine phosphatase-like protein (anti-IA-2), zinc transporter autoantibodies; or an insulin autoantibody (IAA). Please note: A subject who is positive for IAA and negative for the other autoantibodies will not be eligible if the subject has been using insulin for a total of ≥7 days.
* Currently requires insulin for T1DM treatment, or has required insulin therapy (for at least 7 days) for diabetes at some time between the date of diagnosis and the first dose of study drug. Note: subjects currently taking twice daily commercially available pre-mixed insulin will not be eligible.
* MinimalHLA I A and B mismatch and at least one HLA DR match

Exclusion Criteria:

* Body mass index (BMI) ≥ 32.0 kg/m2 or patient weight ≤50kg
* Insulin requirement of >1.0 IU/kg/day
* HbA1c >10%
* Blood Pressure: SBP >160 mmHg or DBP >100 mmHg.
* Chronic disease apart from diabetes, including type 2 diabetes
* Moderate to severe renal impairment as per calculated creatinine clearance (CLcr) < 90 mL/min according to the Cockcroft-Gault formula (Cockcroft-Gault , 1976)
* Presence or history of macroalbuminuria (>300mg/g creatinine).
* Hepatic dysfunction defined by increased ALT/AST upper limit of normal (ULN) and increased total bilirubin > 3 mg/dL [>51.3 μmol/L]
* Pregnant or breast feeding women. Unwillingness to use effective contraceptive measures up to 4 months after the end of study drug administration (females and males)
* Active infection including hepatitis B, hepatitis C, HIV, or tuberculosis (TB) as determined by a positive skin test or clinical presentation, or under treatment for suspected TB. Positive tests are acceptable only if associated with a history of previous vaccination in the absence of any sign of active infection. Positive tests are otherwise not acceptable, even in the absence of any active infection at the time of evaluation.
* Negative screen for Epstein-Barr Virus (EBV) by IgG determination
* Invasive aspergillus, histoplasmosis, or coccidioidomycosis infection within one year prior to study enrollment
* Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin
* Known active alcohol or substance abuse
* Baseline Hb below the lower limits of normal at the local laboratory; lymphopenia (<1,000/µL), neutropenia (<1,500/µL), or thrombocytopenia (platelets <100,000/µL). Participants with lymphopenia are allowed if the investigator determines there is no additional risk and obtains clearance from a hematologist
* A history of Factor V deficiency
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy (e.g., warfarin) after transplantation (low-dose aspirin treatment is allowed) or patients with an international normalized ratio (INR) >1.5
* Severe co-existing cardiac disease, characterized by any one of these conditions:

  * a) recent myocardial infarction (within past 6 months)
  * b) evidence of ischemia on functional cardiac exam within the last year
  * c) left ventricular ejection fraction <30%.
* Symptomatic cholecystolithiasis.
* Acute or chronic pancreatitis.
* Symptomatic peptic ulcer disease.
* Severe unremitting diarrhea, vomiting or other gastrointestinal disorders potentially interfering with the ability to absorb oral medications
* Hyperlipidemia despite medical therapy (fasting low-density lipoprotein [LDL] cholesterol >130 mg/dL, treated or untreated; and/or fasting triglycerides >200 mg/dL)
* Receiving treatment for a medical condition requiring chronic use of systemic steroids, except for the use of ≥ 5 mg prednisone daily, or an equivalent dose of hydrocortisone, for physiological replacement only.
* Treatment with any anti-diabetic medication other than insulin within 4 weeks of enrollment
* Use of any investigational agents within 4 weeks of enrollment.
* Administration of live attenuated vaccine(s) within 2 months of enrollment.
* Any medical condition that, in the opinion of the investigator, will interfere with safe participation in the trial.
* Treatment with any immunosuppressive regimen at the time of enrollment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
plasma C-peptide AUC (mixed meal tolerance test [MMTT]) | 52 weeks
  Mean change from baseline of stimulated plasma C-peptide AUC (mixed meal tolerance test [MMTT])
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 52 weeks

SECONDARY OUTCOMES:
plasma C-peptide AUC (MMTT) | 4,12, 26 weeks and 18, 24, 36, 48, 60 months
  Mean change from baseline in stimulated plasma C-peptide AUC (MMTT) at week 4, 12, 26 and month 18, 24, 36, 48, 60
stimulated plasma C-peptide | 4,12, 26 weeks and 12, 18, 24, 36, 48, 60 months
  Maximum stimulated plasma C-peptide (the highest value at any time point during the MMTT after the mixed meal injection) at baseline, week 4, week 12, week 26 and week 52 and month 18, 24, 36, 48, 60
glucagon AUC (MMTT) | 4,12, 26, 52 weeks
  Mean change from baseline in glucagon AUC (MMTT) at week 4, week 12, week 26 and week 52
HbA1c | 4,12, 26 weeks and 12, 18, 24, 36, 48, 60 months
  Change from baseline in HbA1c at week 52 and HbA1c over time
daily insulin dose | 4,12, 26 weeks and 12, 18, 24, 36, 48, 60 months
  Change from baseline in mean daily insulin dose for the 3 days preceding the visit at weeks 4, 12, 26, 52 and month 18, 24, 36, 48, 60. The mean daily insulin dose value will be calculated, in units of U/kg/day, as the mean of the values of amount of insulin used per day on each of the 3 consecutive days.
hypoglycaemic events | 4,12, 26 weeks and 12, 18, 24, 36, 48, 60 months
  Number of hypoglycaemic events with confirmed self plasma glucose monitoring <3.1 mmol/L (<56 mg/dL) and/or requiring 3rd party intervention (i.e., severe, documented symptomatic and asymptomatic hypoglycaemic events) overall and in 3 monthly intervals
72-hour Continuous Glucose Monitoring | 26 and 52 weeks and 24, 36, 48, 60 months
  Time spent with a plasma glucose <3.9 mmol/L, between 3.9 and 10.0 mmol/L, and >10.0 mmol/L, respectively as performed by 72-hour CGM at baseline, week 26, week 52 and month 24, 36, 48, 60

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Piemonti, MD, Principal Investigator — IRCCS Ospedale San Raffaele; Emanuele Bosi, MD, Study Chair — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy

REFERENCES:
- [Derived] Piemonti L, Bolla AM, Caretto A, Melzi R, Mercalli A, Sordi V, Monti P, Magistretti P, Lampasona V, Marzinotto I, Maffi P, Ramondetta M, Cagni N, Pedone E, Catarinella D, Cardillo M, Caldara R, Bosi E. Induction of immune education in type 1 diabetes through controlled allogeneic islet rejection at onset: a monocentric open-label pilot study. EClinicalMedicine. 2025 Dec 4;90:103685. doi: 10.1016/j.eclinm.2025.103685. eCollection 2025 Dec. PMID 41438972